CLINICAL TRIAL: NCT04412655
Title: International Study on Acute Coronary Syndromes - ST-segment Elevation Myocardial Infarction COVID 19
Brief Title: Primary Angioplasty for STEMI During COVID-19 Pandemic (ISACS-STEMI COVID-19) Registry
Acronym: ISACS-STEMI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Sponsor
Other Study IDs: 115/20
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: ST Elevated Myocardial Infarction Undergoing Mechanical Reperfusion
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI patients treated in March April 2019: Patients with STEMI undergoing mecahnical revascularization from 1th March to 30th April 2019
  Interventions: Device: Percutaneous Coronary Revascularization for STEMI
- STEMI patients treated in March April 2020: Patients with STEMI undergoing mecahnical revascularization from 1th March to 30th April 2020
  Interventions: Device: Percutaneous Coronary Revascularization for STEMI

INTERVENTIONS:
Device: Percutaneous Coronary Revascularization for STEMI — Percutaneous Mechanical Reperfusion for STEMI
  Other Names: Primary angioplasty

SUMMARY:
The ISACS STEMI COVID-19 has been established in response to the emerging outbreak of COVID-19 to provide a European overview to estimate the real impact of COVID-19 pandemic on treatment and outcome of STEMI by primary angioplasty, and to identify any potential category of patients at risk for delay to treatment or no presentation.

DETAILED DESCRIPTION:
This is a retrospective multicenter registry including at least 40 European primary PCI centers with > 120 primary PCI/year (with expected average > 10/month), with the case load of STEMI not expected to be affected by a potential planned reorganization of the STEMI network. The inclusion period will be of 2 months (from March 1st until April 30th). The data will be compared with those retrospectively collected in the same time window of 2019.

Inclusion criteria: STEMI treated by primary angioplasty. Primary study outcome: Number of STEMI patients undergoing primary angioplasty. Secondary study outcomes: Ischemia time and the number of late presenters (> 12 hours from symptoms onset); 3) Door-to-balloon time and the number of patients with a DTB > 30 minutes); 4) In-Hospital mortality.

Data Collection: Data will be collected anonymized through a dedicated CRF. Each center will identify a local Principal Investigator. We will collect information on the study center, demographic, clinical, procedural data. Furthermore, we will collect data on total ischemia time, door-to-balloon time, type of access to the emergency system, COVID positivity, PCI procedure, data on in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria: STEMI Patients undergoing mechanical reperfusion

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI Patients undergoing mechanical reperfusion
Sampling Method: Non-Probability Sample
Enrollment: 6609 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients undergoing primary angioplasty | March April 2019 and 2020
  Number of patients undergoing primary angioplasty
Number of patients undergoing primary angioplasty later than 12 hours from symptoms onset; | March April 2019 and 2020
  Number of patients undergoing primary angioplasty later 12 hours from symptoms onset;
Number of patients undergoing primary angioplasty later than 30 minutes from PCI hospital admission | March April 2019 and 2020
  Number of patients undergoing primary angioplasty later than 30 minutes from PCI hospital admission
In-hospital mortality | March April 2019 and 2020
  In-Hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe De Luca, Novara, Italy

REFERENCES:
- [Derived] De Luca G, Nardin M, Algowhary M, Uguz B, Oliveira DC, Ganyukov V, Zimbakov Z, Cercek M, Okkels Jensen L, Loh PH, Calmac L, Roura Ferrer G, Quadros A, Milewski M, Scotto di Uccio F, von Birgelen C, Versaci F, Ten Berg J, Casella G, Wong Sung Lung A, Kala P, Diez Gil JL, Carrillo X, Dirksen M, Becerra-Munoz VM, Lee MK, Arifa Juzar D, de Moura Joaquim R, Paladino R, Milicic D, Davlouros P, Bakraceski N, Zilio F, Donazzan L, Kraaijeveld A, Galasso G, Lux A, Marinucci L, Guiducci V, Menichelli M, Scoccia A, Yamac AH, Ugur Mert K, Flores Rios X, Kovarnik T, Kidawa M, Moreu J, Flavien V, Fabris E, Martinez-Luengas IL, Boccalatte M, Bosa Ojeda F, Arellano-Serrano C, Caiazzo G, Cirrincione G, Kao HL, Sanchis Fores J, Vignali L, Pereira H, Manzo S, Ordonez S, Ozkan AA, Scheller B, Lehtola H, Teles R, Mantis C, Antti Y, Brum Silveira JA, Zoni R, Bessonov I, Savonitto S, Kochiadakis G, Alexopoulos D, Uribe CE, Kanakakis J, Faurie B, Gabrielli G, Gutierrez Barrios A, Bachini JP, Rocha A, Tam FC, Rodriguez A, Lukito AA, Saint-Joy V, Pessah G, Tuccillo A, Cortese G, Parodi G, Bouraghda MA, Kedhi E, Lamelas P, Suryapranata H, Verdoia M. Impact of chronic obstructive pulmonary disease on short-term outcome in patients with ST-elevation myocardial infarction during COVID-19 pandemic: insights from the international multicenter ISACS-STEMI registry. Respir Res. 2022 Aug 15;23(1):207. doi: 10.1186/s12931-022-02128-0. PMID 35971173
- [Derived] De Luca G, Nardin M, Algowhary M, Uguz B, Oliveira DC, Ganyukov V, Zimbakov Z, Cercek M, Jensen LO, Loh PH, Calmac L, Roura Ferrer G, Quadros A, Milewski M, Scotto di Uccio F, von Birgelen C, Versaci F, Ten Berg J, Casella G, Lung AWS, Kala P, Diez Gil JL, Carrillo X, Dirksen M, Becerra-Munoz VM, Lee MK, Juzar DA, de Moura Joaquim R, Paladino R, Milicic D, Davlouros P, Bakraceski N, Zilio F, Donazzan L, Kraaijeveld A, Galasso G, Lux A, Marinucci L, Guiducci V, Menichelli M, Scoccia A, Yamac AH, Mert KU, Flores Rios X, Kovarnik T, Kidawa M, Moreu J, Flavien V, Fabris E, Martinez-Luengas IL, Boccalatte M, Bosa Ojeda F, Arellano-Serrano C, Caiazzo G, Cirrincione G, Kao HL, Sanchis Fores J, Vignali L, Pereira H, Manzo S, Ordonez S, Arat Ozkan A, Scheller B, Lehtola H, Teles R, Mantis C, Antti Y, Brum Silveira JA, Zoni R, Bessonov I, Savonitto S, Kochiadakis G, Alexopulos D, Uribe CE, Kanakakis J, Faurie B, Gabrielli G, Gutierrez Barrios A, Bachini JP, Rocha A, Tam FC, Rodriguez A, Lukito AA, Saint-Joy V, Pessah G, Tuccillo A, Cortese G, Parodi G, Bouraghda MA, Kedhi E, Lamelas P, Suryapranata H, Verdoia M. Renin-angiotensin system inhibitors and mortality among diabetic patients with STEMI undergoing mechanical reperfusion during the COVID-19 pandemic. Diabet Epidemiol Manag. 2021 Oct-Dec;4:100022. doi: 10.1016/j.deman.2021.100022. Epub 2021 Oct 30. PMID 35072135
- [Derived] De Luca G, Algowhary M, Uguz B, Oliveira DC, Ganyukov V, Zimbakov Z, Cercek M, Jensen LO, Loh PH, Calmac L, Roura-Ferrer G, Quadros A, Milewski M, Scotto di Uccio F, von Birgelen C, Versaci F, Ten Berg J, Casella G, Wong ASL, Kala P, Diez Gil JL, Carrillo X, Dirksen MT, Becerra-Munoz VM, Kang-Yin Lee M, Juzar DA, de Moura Joaquim R, Paladino R, Milicic D, Davlouros P, Bakraceski N, Zilio F, Donazzan L, Kraaijeveld AO, Galasso G, Lux A, Marinucci L, Guiducci V, Menichelli M, Scoccia A, Yamac A, Ugur Mert K, Flores Rios X, Kovarnik T, Kidawa M, Moreu J, Flavien V, Fabris E, Lozano Martinez-Luengas I, Boccalatte M, Bosa Ojeda F, Arellano-Serrano C, Caiazzo G, Cirrincione G, Kao HL, Sanchis Fores J, Vignali L, Pereira H, Manzo-Silberman S, Ordonez S, Ozkan AA, Scheller B, Lehtola H, Teles R, Mantis C, Ylitalo A, Brum Silveira JA, Zoni R, Bessonov I, Savonitto S, Kochiadakis G, Alexopoulos D, Uribe C, Kanakakis J, Faurie B, Gabrielli G, Gutierrez A, Bachini JP, Rocha A, Tam FC, Rodriguez A, Lukito A, Saint-Joy V, Pessah G, Tuccillo B, Cortese G, Parodi G, Bouraghda MA, Kedhi E, Lamelas P, Suryapranata H, Nardin M, Verdoia M; ISACS-STEMI COVID-19; Collaborators. COVID-19 pandemic, mechanical reperfusion and 30-day mortality in ST elevation myocardial infarction. Heart. 2022 Mar;108(6):458-466. doi: 10.1136/heartjnl-2021-319750. Epub 2021 Oct 28. PMID 34711661
- [Derived] De Luca G, Debel N, Cercek M, Jensen LO, Vavlukis M, Calmac L, Johnson T, Ferrer GR, Ganyukov V, Wojakowski W, Kinnaird T, von Birgelen C, Cottin Y, IJsselmuiden A, Tuccillo B, Versaci F, Royaards KJ, Berg JT, Laine M, Dirksen M, Siviglia M, Casella G, Kala P, Diez Gil JL, Banning A, Becerra V, De Simone C, Santucci A, Carrillo X, Scoccia A, Amoroso G, Van't Hof AW, Kovarnik T, Tsigkas G, Mehilli J, Gabrielli G, Rios XF, Bakraceski N, Levesque S, Cirrincione G, Guiducci V, Kidawa M, Spedicato L, Marinucci L, Ludman P, Zilio F, Galasso G, Fabris E, Menichelli M, Garcia-Touchard A, Manzo S, Caiazzo G, Moreu J, Fores JS, Donazzan L, Vignali L, Teles R, Benit E, Agostoni P, Ojeda FB, Lehtola H, Camacho-Freiere S, Kraaijeveld A, Antti Y, Boccalatte M, Deharo P, Martinez-Luengas IL, Scheller B, Varytimiadi E, Moreno R, Uccello G, Faurie B, Gutierrez Barrios A, Milewski M, Bruwiere E, Smits P, Wilbert B, Di Uccio FS, Parodi G, Kedhi E, Verdoia M. Impact of SARS-CoV-2 positivity on clinical outcome among STEMI patients undergoing mechanical reperfusion: Insights from the ISACS STEMI COVID 19 registry. Atherosclerosis. 2021 Sep;332:48-54. doi: 10.1016/j.atherosclerosis.2021.06.926. Epub 2021 Jul 21. PMID 34391035
- [Derived] De Luca G, Cercek M, Jensen LO, Vavlukis M, Calmac L, Johnson T, Roura I Ferrer G, Ganyukov V, Wojakowski W, von Birgelen C, Versaci F, Ten Berg J, Laine M, Dirksen M, Casella G, Kala P, Diez Gil JL, Becerra V, De Simone C, Carrill X, Scoccia A, Lux A, Kovarnik T, Davlouros P, Gabrielli G, Flores Rios X, Bakraceski N, Levesque S, Guiducci V, Kidawa M, Marinucci L, Zilio F, Galasso G, Fabris E, Menichelli M, Manzo S, Caiazzo G, Moreu J, Sanchis Fores J, Donazzan L, Vignali L, Teles R, Bosa Ojeda F, Lehtola H, Camacho-Freiere S, Kraaijeveld A, Antti Y, Boccalatte M, Martinez-Luengas IL, Scheller B, Alexopoulos D, Uccello G, Faurie B, Gutierrez Barrios A, Wilbert B, Cortese G, Moreno R, Parodi G, Kedhi E, Verdoia M. Impact of COVID-19 pandemic and diabetes on mechanical reperfusion in patients with STEMI: insights from the ISACS STEMI COVID 19 Registry. Cardiovasc Diabetol. 2020 Dec 18;19(1):215. doi: 10.1186/s12933-020-01196-0. PMID 33339541
- [Derived] De Luca G, Verdoia M, Cercek M, Jensen LO, Vavlukis M, Calmac L, Johnson T, Ferrer GR, Ganyukov V, Wojakowski W, Kinnaird T, van Birgelen C, Cottin Y, IJsselmuiden A, Tuccillo B, Versaci F, Royaards KJ, Berg JT, Laine M, Dirksen M, Siviglia M, Casella G, Kala P, Diez Gil JL, Banning A, Becerra V, De Simone C, Santucci A, Carrillo X, Scoccia A, Amoroso G, Lux A, Kovarnik T, Davlouros P, Mehilli J, Gabrielli G, Rios XF, Bakraceski N, Levesque S, Cirrincione G, Guiducci V, Kidawa M, Spedicato L, Marinucci L, Ludman P, Zilio F, Galasso G, Fabris E, Menichelli M, Garcia-Touchard A, Manzo S, Caiazzo G, Moreu J, Fores JS, Donazzan L, Vignali L, Teles R, Benit E, Agostoni P, Bosa Ojeda F, Lehtola H, Camacho-Freiere S, Kraaijeveld A, Antti Y, Boccalatte M, Deharo P, Martinez-Luengas IL, Scheller B, Alexopoulos D, Moreno R, Kedhi E, Uccello G, Faurie B, Gutierrez Barrios A, Di Uccio FS, Wilbert B, Smits P, Cortese G, Parodi G, Dudek D. Impact of COVID-19 Pandemic on Mechanical Reperfusion for Patients With STEMI. J Am Coll Cardiol. 2020 Nov 17;76(20):2321-2330. doi: 10.1016/j.jacc.2020.09.546. PMID 33183506